CLINICAL TRIAL: NCT06556368
Title: A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Three-arm Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal Tarcocimab Tedromer and Tabirafusp Tedromer Compared With Intravitreal Aflibercept in Participants With Neovascular (Wet) Age-related Macular Degeneration (wAMD)
Brief Title: A Study to Evaluate the Efficacy and Safety of Tarcocimab Tedromer and Tabirafusp Tedromer Compared to Aflibercept in Participants With Neovascular (Wet) Age-related Macular Degeneration (wAMD) - DAYBREAK
Acronym: DAYBREAK
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS301P109
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-03

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Wet AMD; KSI-301; KSI-501; Tarcocimab; Tabirafusp; Aflibercept; Antibody biopolymer conjugate; AMD; Anti-VEGF; Vascular endothelial growth factor; Kodiak Sciences
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 into one of three treatment groups: tarcocimab-ted, tabirafusp-ted or aflibercept.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tarcocimab tedromer 5 mg (KSI-301) (Experimental): Intravitreal injection of tarcocimab tedromer once every 4 weeks for 4 monthly doses followed by individualized dosing every 4 to 24 weeks.
  Interventions: Drug: Tarcocimab tedromer
- Tabirafusp tedromer 5 mg (KSI-501) (Experimental): Intravitreal injection of tabirafusp tedromer once every 4 weeks for 4 monthly doses followed by every-8-week dosing with additional individualized dosing (up to monthly dosing)
  Interventions: Drug: Tabirafusp tedromer
- Aflibercept 2 mg (Active Comparator): Intravitreal injection of aflibercept once every 4 weeks for 3 monthly doses followed by every-8-week dosing
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Tarcocimab tedromer — Intravitreal injection
  Other Names: KSI-301
  Arms: Tarcocimab tedromer 5 mg (KSI-301)
Drug: Tabirafusp tedromer — Intravitreal injection
  Other Names: KSI-501
  Arms: Tabirafusp tedromer 5 mg (KSI-501)
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
A Study to Evaluate the Efficacy and Safety of Tarcocimab Tedromer and Tabirafusp Tedromer Compared to Aflibercept in Participants with Neovascular (Wet) Age-related Macular Degeneration (wAMD)

ELIGIBILITY:
Inclusion Criteria:

* Active, treatment-naïve choroidal neovascularization (CNV) secondary to AMD, including subfoveal, juxtafoveal, and extrafoveal lesions, or retinal angiomatous proliferations (RAP) lesions with a CNV component that affects the central subfield, as evidenced by FA or OCT in the Study Eye at Screening
* BCVA ETDRS score between 78 and 25 letters (Snellen equivalent ~20/32 and 20/320) inclusive, in the Study Eye at screening and reconfirmed at Day 1.
* Capable of giving signed informed consent.

Exclusion Criteria:

* BCVA of hand motion or worse in the non-Study Eye or non-physical presence of a non-Study Eye (i.e., monocular)
* Fibrosis or atrophy of >50% of the lesion size and/or involving the foveal center of the Study Eye at Screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | Week 48
  Mean change in BCVA from Day 1 to Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (72):
- United States (71):
  - Associated Retina Consultants, Gilbert, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Retina Associates SW, Tucson, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Global Research Management, Inc. - Lugene Eye Institute, Glendale, California
  - Retinal Consultants Medical Group, Inc., Modesto, California
  - California Eye Specialists Medical Group, Inc., Pasadena, California
  - California Eye Specialists Medical Group, Inc., Redlands, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Retina Group of New England, PC, Waterford, Connecticut
  - Blue Ocean Clinical Research, Clearwater, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Retina Group of Florida, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Retina Associates, Ltd, Elmhurst, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Associated Vitreoretinal and Uveitis Consultants LLC, Carmel, Indiana
  - Midwest Eye Institute, Carmel, Indiana
  - The Retina Care Center, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Minnesota, Edina, Minnesota
  - Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - Mississippi Retina Associates, Madison, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Retina Consultants of Nevada, Henderson, Nevada
  - Long Island Vitreoretinal Consultants, Hauppauge, New York
  - Retina Vitreous Surgeons of CNY PC, Liverpool, New York
  - Retina Associates of Western NY, Rochester, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - North Carolina Retina Associates, Cary, North Carolina
  - Piedmont Retina Specialist, Greensboro, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Western Carolina Clinical Research, LLC, Winston-Salem, North Carolina
  - Retina Northwest, Portland, Oregon
  - Cascade Medical Research Institute, Springfield, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Vision Research Solutions PLLC, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Aiken, South Carolina
  - Charleston Neuroscience Institute, LLC, Beaufort, South Carolina
  - Charleston Neuroscience Institute, LLC, Charleston, South Carolina
  - Charleston Neuroscience Institute, LLC, Ladson, South Carolina
  - Charleston Neuroscience Institute, Mt. Pleasant, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Ophthalmology Ltd, Sioux Falls, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Panhandle Eye Group, LLP. - Southwest Retina Specialists, Amarillo, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, PLLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Star Vision Research, Burleson, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Texas Retina Center, Houston, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates, PLLC, Round Rock, Texas
  - Retinal Consultants of Houston dba Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, Schertz, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Pacific Northwest Retina, Bellevue, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - Eye Clinic of Wisconsin, Wausau, Wisconsin
- Emanuelli Research & Development Center, LLC, Arecibo, Puerto Rico, Puerto Rico